CLINICAL TRIAL: NCT01904123
Title: A Phase I Trial of WP1066 in Patients With Recurrent Malignant Glioma and Brain Metastasis From Melanoma
Brief Title: STAT3 Inhibitor WP1066 in Treating Patients With Recurrent Malignant Glioma or Progressive Metastatic Melanoma in the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0358; NCI-2015-00163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0358 (Other: M D Anderson Cancer Center); P50CA127001 (NIH); P50CA093459 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Recurrent Brain Neoplasm; Recurrent Glioblastoma; Recurrent Malignant Glioma
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Glioblastoma; Glioma | interventions — WP1066

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (STAT3 inhibitor WP1066) (Experimental): Patients receive STAT3 inhibitor WP1066 PO BID on Monday, Wednesday, and Friday of weeks 1 and 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: STAT3 Inhibitor WP1066

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: STAT3 Inhibitor WP1066 — Given PO
  Other Names: WP1066

SUMMARY:
This phase I trial studies the side effects and best dose of STAT3 inhibitor WP1066 in treating patients with malignant glioma that has come back or melanoma that has spread to the brain and is growing, spreading, or getting worse. STAT3 inhibitor WP1066 may stop the growth of tumor cells and modulate the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. Identify the maximum tolerated dose (MTD) of STAT3 inhibitor WP1066 (WP1066) in patients with recurrent malignant glioma (glioblastoma, anaplastic glioma), and melanoma patients with progressive brain metastasis.

II. Assess the safety and tolerability of WP1066 in patients with recurrent malignant glioma and melanoma patients with progressive brain metastasis using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) with special attention directed at determining whether any induced autoimmune reactions occur.

SECONDARY OBJECTIVES:

I. Pharmacokinetic analysis of the in vivo bioavailability of WP1066. II. Assess overall response rate (ORR) in patients with recurrent malignant gliomas and progressive metastatic melanoma to the brain.

III. Assess immunological response in patients with recurrent malignant glioma and melanoma patients with progressive brain metastasis treated with WP1066.

IV. Assess time to radiographically assessed progression and/or response in patients treated with WP1066.

V. Assess progression-free survival (PFS) and overall survival (OS) in patients treated with WP1066.

VI. Estimate the proportion of patients treated with WP1066 who develop additional melanoma metastatic lesions, including those in the central nervous system (CNS).

OUTLINE: This is a dose-escalation study.

Patients receive STAT3 inhibitor WP1066 orally (PO) twice daily (BID) on Monday, Wednesday, and Friday of weeks 1 and 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed progressive brain metastases from melanoma or recurrent/progressive malignant glioma (glioblastoma, anaplastic glioma), for which standard curative or palliative measures, with the exception of surgery, do not exist or are no longer effective
* Patients must have measurable disease in the brain, defined as at least one lesion that can be accurately measured in at least one dimension as >= 10 mm by brain magnetic resonance imaging (MRI); MRI of the brain (with and without gadolinium enhancement) is to be performed using standard 5-mm slices with 2.5-mm spacing for comparison to subsequent MRI scans
* In the case of malignant glioma patients, they must have previously undergone standard-of-care treatment including surgery, radiation, and first line adjuvant chemotherapy prior to the experimental treatment (WP1066); in the case of melanoma patients with brain metastasis, they may have previously undergone a resection (with radiographic evidence of progression), have undergone gamma knife radiosurgery (with radiographic evidence of progression), or have been treated with other systemic therapies that failed
* Karnofsky performance scale score >= 60%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.6
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT)/partial thromboplastin time (PTT) < 1.5 x normal institutional standard
* Ability to understand and the willingness to sign a written informed consent document
* Melanoma patients must be intolerant of, or have disease that has proven refractory to approved therapies such as BRAF or MEK inhibitors for BRAF-positive metastatic melanoma and/or checkpoint blockade with either anti-PD1 or anti-CTLA-4 for metastatic melanoma
* Willing and able to tolerate brain MRI's with contrast
* Patients with stable seizures (e.g., no seizures for >= 14 days and not requiring escalation or addition of anti-epileptic drugs for 14 days from starting treatment) will be eligible
* Patients who are eligible for the surgical expansion cohort are identified by the clinical team who have made the independent decision that the patient would benefit from non-emergent palliative surgical resection (i.e. they are not a candidate for gamma knife or other type of standard therapy)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; biological agents, immune modulators, and targeted therapeutic approaches require a 2-week washout window
* Patients who are receiving any other investigational agents require a 4 week washout period; patients who have received cellular or gene therapy at any time are not eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to WP1066
* The enzymatic metabolism profile of WP1066 is unknown; patients who are receiving drugs that significantly interact with the cytochrome P450 (CYP450) enzyme(s) are ineligible; however, if they are switched to other medications with a 2-week washout window, they will be eligible; patients are also excluded if they have been exposed within 7 days of planned first study treatment day to medications that are predominantly cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6), cytochrome P450, family 2, subfamily C, polypeptide 9 (2C9) or cytochrome P450, family 2, subfamily C, polypeptide 19 (2C19) substrates, strong inhibitors or inducers, and sensitive substrates of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) with narrow therapeutic range; patients requiring escalation of the corticosteroid dose will be excluded, but patients receiving a stable or decreasing dose for at least one week will be eligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No single lesion can be larger than 3 cm in maximal diameter; there may not be midline shift exceeding 5 mm or hydrocephalus
* Pregnant women are excluded from this study because WP1066 could potentially be teratogenic or have abortifacient effects; breastfeeding should be discontinued if the mother is treated with WP0166; female subjects of childbearing potential should be willing to use 2 methods of birth control prior to study entry, during the study, and for 2 months after the last dose of the study drug or be surgically sterile; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of WP1066 administration
* Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with WP1066
* Patients who have received bevacizumab, Gliadel, or are on active therapy with Optune are not eligible
* The potential for further hemorrhaging with the use of WP1066 is unknown; furthermore, because brain melanoma metastases commonly hemorrhage, toxicity may be inappropriately attributed to WP1066 in this setting; it will be at the principal investigator's (PIs) discretion to enroll a patient who has a small, asymptomatic brain hemorrhage, but patients who have had symptomatic hemorrhages will be excluded
* Patients with uncontrolled seizures or seizure requiring escalation or addition of anti-epileptic drugs will be excluded
* Because one of the secondary objectives is PFS based on radiographic volumetric analysis of the tumor, the presence of diffuse leptomeningeal disease will be an exclusion criterion for this study; this is secondary to the inadequacy of measuring the extent of the tumor burden within this setting and the very poor prognosis of these patients
* The cardiac toxicities of WP1066 are unknown; thus, patients who have a corrected QT (QTc) interval > 450 ms at base line will be excluded; concomitant use of agents that prolong the QT interval will be avoided
* Malignant glioma patients within 12 weeks of completion of radiation concurrent temozolomide will be excluded
* Melanoma patients with large or symptomatic brain metastasis, and in whom neurosurgical removal is indicated will not be eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of JAK2 inhibitor WP1066, defined as the dose level at which 0/6 or 1/6 patients experience a dose limiting toxicity (DLT) with at least 2 patients experiencing DLT at the next higher dose level | 28 days
  A DLT will be defined as an adverse event or an abnormal laboratory value assessed as being at least possibly related to the investigation agent that occurs during the first 28 days after administration of the first dose of JAK2 inhibitor WP1066 and will be assigned a grade based on National Cancer Institute (NCI) Common Terminology Criteria (CTC). Any grade toxicity at least possibly related to WP1066 that leads to dose delay of >= 2 weeks will be considered a DLT.
Incidence of adverse events assessed using NCI CTC | Up to 2 months after the last study drug dose

SECONDARY OUTCOMES:
Pharmacokinetic analysis of the in vivo bioavailability of JAK2 inhibitor WP1066 | Days 1, 2, 14, and 15 of course 1
Proportion of patients reaching complete response or partial response | Up to 2 months after the last study drug dose
  Estimated with a 95% confidence interval.
Duration of response | Up to 2 months after the last study drug dose
  Estimated using Kaplan-Meier survival curves. Cox proportional hazards regression methodology may be used to assess the association between duration of response or survival and clinical and demographic characteristics of interest.
Overall survival | Up to 2 months after the last study drug dose
  Estimated using Kaplan-Meier survival curves. Cox proportional hazards regression methodology may be used to assess the association between duration of response or survival and clinical and demographic characteristics of interest.
Progression free survival | Up to 2 months after the last study drug dose
  Estimated using Kaplan-Meier survival curves. Cox proportional hazards regression methodology may be used to assess the association between duration of response or survival and clinical and demographic characteristics of interest.
The proportion of patients who develop additional melanoma metastatic lesions | Up to 2 months after the last study drug dose
  Estimated with a 95% confidence interval.
Change in regulatory T cell numbers | Baseline up to 2 months after the last study drug dose
  Tested using paired t-tests or Wilcoxon signed-rank tests, as appropriate. The longitudinal analysis for all markers will be similar using generalized linear mixed-effects (GLMM) models to assess the significance of the changing values over time and estimating the trajectory.
Change in the number of peripheral blood mononuclear cells expressing phosphorylated STAT3 | Baseline up to 2 months after the last study drug dose
  Tested using paired t-tests or Wilcoxon signed-rank tests, as appropriate. The longitudinal analysis for all markers will be similar using GLMM models to assess the significance of the changing values over time and estimating the trajectory.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Heimberger, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Choi HK, Park SH, Lee J, Hwang JT. Review of Patents for Anticancer Agents Targeting Adenosine Monophosphate-Activated Protein Kinase. J Med Food. 2023 Sep;26(9):605-615. doi: 10.1089/jmf.2023.K.0026. Epub 2023 Aug 16. PMID 37590001
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org